CLINICAL TRIAL: NCT00118053
Title: A Phase II Trial of Taxotere, Carboplatin and Herceptin in Locally Advanced or Inflammatory Breast Cancer
Brief Title: Trastuzumab, Docetaxel, and Carboplatin in Treating Women With Stage II, Stage III, or Inflammatory Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040412;CDR0000433511; P30CA072720 (NIH); CINJ-040412 (Other: Cancer Institute of New Jersey); 0220045191 (Other: UMDNJ-RWJMS IRB); CINJ-NJ1104 (Other: Cancer Institute of New Jersey)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-09

CONDITIONS: Breast Cancer
Keywords: inflammatory breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Trastuzumab; Carboplatin; Docetaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Docetaxel, Carboplatin and Trastuzumab (Experimental): A total of six cycles of TCH [(Taxotere® (75 mg/m2) + Carboplatin (AUC = 6) + Herceptin® (2 mg/kg weekly after a 4 mg/kg load on Day 1)] will be administered every 3 weeks.Three weeks after receiving the sixth cycle of TCH, all patients will be restaged.
  * Those determined to have localized and operable disease (as determined by surgical consultation) will undergo a modified radical mastectomy or lumpectomy and axillary node dissection. After recovery from surgery, the patients will receive whole breast or chest wall irradiation (as determined by radiologist) with concurrent Herceptin® (6 mg/kg). Following radiation, patients will continue Herceptin® (6 mg/kg) every 3 weeks until they have been on study for a total of 52 weeks.
  * If patients are staged and are negative they will continue Herceptin® (6 mg/kg)every 3 weeks until they have been on study for a total of 52 weeks.
  Interventions: Biological: herceptin; Drug: carboplatin; Drug: docetaxel; Procedure: conventional surgery; Procedure: radiation therapy

INTERVENTIONS:
Biological: herceptin
  Other Names: trastuzumb
Drug: carboplatin
Drug: docetaxel
  Other Names: Taxotere
Procedure: conventional surgery — Modified radical mastectomy or lumpectomy and axillary node dissection
Procedure: radiation therapy — Whole breast or chest wall irradiation (as determined by radiologist)

SUMMARY:
RATIONALE: Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as docetaxel and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving trastuzumab together with docetaxel and carboplatin may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving trastuzumab together with docetaxel and carboplatin works in treating women with stage II, stage III, or inflammatory breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the antitumor activity of trastuzumab (Herceptin^®), docetaxel, and carboplatin, as measured by tumor response rate, in women with previously untreated HER2/neu-positive stage IIB, IIIA, IIIB, or IIIC or inflammatory breast cancer.

Secondary

* Determine the pathological complete response in patients treated with this regimen.
* Determine the disease-free survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine pathologic and molecular markers for predicting efficacy of this regimen in these patients.

OUTLINE: This is a non-randomized, multicenter study.

* Course 1 (days 1-28): Patients receive trastuzumab (Herceptin^®) IV over 30-90 minutes on days 1, 8, 15, and 22 and docetaxel IV over 1 hour and carboplatin IV over 30-60 minutes on day 8.
* Course 2-6: Patients receive trastuzumab IV over 30 minutes on days 1, 8, and 15 during courses 2-5 and on days 1, 8, 15, and 22 during course 6. Patients also receive docetaxel IV over 1 hour and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 5 additional courses (6 courses total) in the absence of disease progression or unacceptable toxicity.

Three weeks after completion of course 6, patients undergo restaging. Patients with local operable disease undergo modified radical mastectomy or lumpectomy and axillary node dissection followed by radiotherapy. Patients also receive trastuzumab IV once every 3 weeks for up to 52 weeks of total treatment (including the 6 courses of trastuzumab, docetaxel, and carboplatin) in the absence of disease progression or unacceptable toxicity. Patients who do not have local operable disease continue to receive trastuzumab as above.

PROJECTED ACCRUAL: A total of 13-43 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer, meeting 1 of the following stage criteria:

  * Stage IIB (T3, N0)
  * Stage IIIA (N0-N2)
  * Stage IIIB (T4, N0-2)
  * Stage IIIC
  * Inflammatory breast cancer
* HER2/neu-positive disease by fluorescence in situ hybridization
* Biopsy-accessible tumor
* Measurable disease by physical examination or x-ray
* No stage IV disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* At least 8 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Meets 1 of the following criteria:

  * SGOT and SGPT ≤ 5 times upper limit of normal (ULN) AND alkaline phosphatase normal
  * SGOT and SGPT ≤ 1.5 times ULN AND alkaline phosphatase ≤ 2.5 times ULN
  * SGOT and SGPT normal AND alkaline phosphatase ≤ 5 times ULN
* Bilirubin normal

Renal

* Creatinine normal
* No pre-existing clinically significant renal disease that is not related to the malignancy

Cardiovascular

* Ejection fraction ≥ 50% by MUGA
* No pre-existing clinically significant cardiac disease that is not related to the malignancy
* No history of congestive heart failure

Pulmonary

* No pre-existing clinically significant pulmonary disease that is not related to the malignancy

Gastrointestinal

* No severe malnutrition
* No intractable emesis

Neurologic

* No pre-existing clinically significant neurologic disease that is not related to the malignancy
* No peripheral neuropathy ≥ grade 2

  * No nerve damage from diabetes

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective non-hormonal contraception during and for 4 weeks after completion of study treatment
* No known allergic reaction to study drugs
* No active infection
* No other malignancy except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No other pre-existing clinically significant disease that is not related to the malignancy
* No other serious or significant medical condition that would preclude study participation
* No other contraindication to study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No other concurrent immunotherapy

Chemotherapy

* No prior chemotherapy for the malignancy
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy for the malignancy

Radiotherapy

* No concurrent radiotherapy

Surgery

* No concurrent surgery for the malignancy

Other

* More than 2 weeks since prior and no concurrent herbal remedies or aspirin-containing products
* No other concurrent investigational or commercial agents or therapies for the malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L. Toppmeyer, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (9):
- United States (9):
  - Central Jersey Oncology Center, PA - East Brunswick, East Brunswick, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Mountainside Hospital Cancer Center, Montclair, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - UMDNJ University Hospital, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://www.clinicaltrials.gov/ct2/show/NCT00118053

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Cancer Institute of New Jersey (a comprehensive cancer center) and 3 community hospitals within NJ from March 2005 through January 2007.
Groups:
- Docetaxel, Carboplatin and Trastuzumab: A total of six cycles of TCH [(Taxotere® (75 mg/m2) + Carboplatin (AUC = 6) + Herceptin® (2 mg/kg weekly after a 4 mg/kg load on Day 1)] will be administered every 3 weeks.Three weeks after receiving the sixth cycle of TCH, all patients will be restaged.
  * Those determined to have localized and operable disease will undergo a modified radical mastectomy or lumpectomy and axillary node dissection. After recovery from surgery, the patients will receive whole breast or chest wall irradiation (as determined by radiologist) with concurrent Herceptin® (6 mg/kg). Following radiation, patients will continue Herceptin® (6 mg/kg) every 3 weeks until they have been on study for a total of 52 weeks.
  * If patients are staged and are negative they will continue Herceptin® (6 mg/kg)every 3 weeks until they have been on study for a total of 52 weeks.
Period: Overall Study
Arm/Group | Docetaxel, Carboplatin and Trastuzumab
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Docetaxel, Carboplatin and Trastuzumab
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Antitumor Activity as Measured by Response Rate
Time Frame: 5 years
Population: Study was terminated early and insufficient data were collected to evaluate this outcome measure.
Arm/Group | Docetaxel, Carboplatin and Trastuzumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Pathological Complete Response
Time Frame: 5 years
Population: Study was terminated early and insufficient data were collected to evaluate this outcome measure.
Arm/Group | Docetaxel, Carboplatin and Trastuzumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Disease-free Survival
Time Frame: 10 years
Population: Study was terminated early and insufficient data were collected to evaluate this outcome measure.
Arm/Group | Docetaxel, Carboplatin and Trastuzumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Pathologic and Molecular Markers for Predicting Efficacy
Time Frame: 5 years
Population: Study was terminated early and insufficient data were collected to evaluate this outcome measure.
Arm/Group | Docetaxel, Carboplatin and Trastuzumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Docetaxel, Carboplatin and Trastuzumab
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel, Carboplatin and Trastuzumab (N=5)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel, Carboplatin and Trastuzumab (N=5)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (7)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2 (3)
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1 (2)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Glucose, serum-high (hyperglycemia) (Investigations) | 2 (6)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (6)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1 (5)
Potassium, serum-low (hypokalemia) (Investigations) | 1 (2)
Sodium, serum-low (hyponatremia) (Investigations) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (4)
Blood/Bone Marrow - Other (Specify, __) (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (3)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (4)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pain - Extremity-limb (General disorders) | 2 (2)
Pain - Abdomen NOS (General disorders) | 1 (1)
Pain - Other (Specify, __) (General disorders) | 1 (1)
Thrombotic microangiopathy (e.g., thrombotic thrombocytopenic purpura [TTP] or hemolytic uremic synd (Vascular disorders) | 1 (2)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (General disorders) | 1 (1)
Infection with unknown ANC - Bladder (urinary) (Infections and infestations) | 1 (1)
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 1 (1)
Edema: limb (Vascular disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 (1)
Neurology - Other (Specify, __) (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (5)
Eyelid dysfunction (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes